CLINICAL TRIAL: NCT06246604
Title: Ultrasound Screening for Asymptomatic Deep Vein Thrombosis in Critically Ill Patient: a Multicenter Trial
Brief Title: Screening for Deep Vein Thrombosis in Intensive Care
Acronym: DVT_ICU2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Of Perugia (Other)
Collaborators: Azienda Ospedaliera di Perugia (Other); Azienda Ospedaliera di Terni (Unknown); Azienda Sanitaria Locale N.1 dell'Umbria (Other); USL Umbria 2 (Unknown)
Responsible Party: Principal Investigator, Stefano Ministrini, Researcher, University Of Perugia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: DVT_ICU2
Record Dates: First submitted 2023-11-26; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Intervention Model Description: Multicenter trial, involving 2 intervention arms: screening and standard-of-care.
  Centers are randomly allocated to provide the screening or the standard-of-care.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Enrolling centers are blinded to each others. Investigators are blinded to centers allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screening (Experimental): Patients will receive an ultrasound screening for DVT between 48 to 96 hours after the admission to the intensive care. In case of negative ultrasound:
  * if the pharmacological thromboprophylaxis is NOT possible, ultrasound is repeated after 48-96 hours;
  * if the pharmacological thromboprophylaxis is possible, re-evaluation is warrant only in case of clinical changes.
  In case of positive ultrasound:
  * if the DVT is proximal, it must be treated according to guidelines. Re-evaluation is warranted only in case of clinical changes;
  * if the DVT is distal and a full or intermediate anti-thrombotic treatment is possible, re-evaluation is warrant only in case of clinical changes;
  * if the DVT is distal and a full or intermediate anti-thrombotic treatment is NOT possible, the ultrasound is repeated after 48-96 hours.
  Interventions: Diagnostic Test: Ultrasound screening for lower limbs DVT
- Standard-of-care (Active Comparator): Ultrasound examination are performed according to clinical risk of DVT
  Interventions: Diagnostic Test: Standard-of-care

INTERVENTIONS:
Diagnostic Test: Ultrasound screening for lower limbs DVT — Using a linear ultrasound probe (7.5-12 MHz) a compression ultrasound of the lower limbs is performed, from the hip to the ankle. The exam is completed by the use of Doppler.
  Arms: Screening
Diagnostic Test: Standard-of-care — Ultrasound examination of lower limbs is performed according to clinical risk of DVT
  Arms: Standard-of-care

SUMMARY:
Background: venous thromboembolism (VTE) is a common complication in critically ill patients, admitted to the Intensive Care Units (ICUs). At the present time, there is no validated score to estimate risks and benefits of antithrombotic pharmacological prophylaxis in this subset of patients. Results of a pilot study showed that ultrasound (US) screening for deep vein thrombosis (DVT) is associated with a reduced incidence of proximal DVT, up front to an overall increased discovery rate of DVTs. The reduced incidence of proximal DVT could be attributed to an early diagnosis of distal and muscular DVTs, which would eventually receive a more adequate management. Proximal DVTs are associated with a worse long-term prognosis than distal or muscular DVTs, so it can be hypothesized that the active US screening could lead to an improvement of in-hospital and long-term prognosis of patients admitted to the ICU.

Aim of the study: to test whether an active US screening may reduce the incidence of proximal DVT and improve the in-hospital and long-term prognosis of patients admitted to the ICU.

Expected relevance: systematic screening for DVT could improve the management of the pharmacological antithrombotic treatment, leading to a reduction of thromboembolic and bleeding complications. This will eventually lead to an improved in-hospital and long-term prognosis.

ELIGIBILITY:
Inclusion Criteria:

* any patient admitted to ICU with a length-of-stay in ICU >96 hours

Exclusion Criteria:

* pregnancy
* SARS-CoV-2 infection
* established DVT or pulmonary embolism at admission
* established coagulation disorder
* presence of inferior vena cava filter at the admission
* admission from the ICU of another hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Proximal deep vein thrombosis | Within 48-72 hours after admission to ICU
  Deep vein thrombosis located above the popliteal area

SECONDARY OUTCOMES:
Mortality in ICU | From admission to ICU until the date of death from any cause or transfer to other facility, assessed up to 30 days
  Death rate during the hospitalization in ICU
In-hospital mortality | From admission to ICU until the date of death from any cause or discharge, assessed up to 30 days
  Death rate during the overall hospital stay
90-day mortality | Within 90 days after the admission of the ICU
  Death rate within 90 days after the admission to the ICU

OTHER OUTCOMES:
Major bleeding | From admission to ICU until the date of death from any cause or transfer to other facility, assessed up to 30 days
  Clinically relevant bleeding
Anemization | From admission to ICU until the date of death from any cause or transfer to other facility, assessed up to 30 days
  Hemoglobin reduction >2 g/dL or need for transfusion during the ICU stay
Pulmonary embolism | From admission to ICU until the date of death from any cause or transfer to other facility, assessed up to 30 days
  Pulmonary embolism diagnosed by chest CT

CONTACTS AND LOCATIONS:
Overall Officials: Leonella Pasqualini, MD, Study Director — University Of Perugia
Locations (5):
- Italy (5):
  - Azienda Sanitaria Locale N.1 dell'Umbria, Città di Castello
  - Azienda Sanitaria Locale N.2 dell'Umbria, Foligno
  - Azienda Sanitaria Locale N.1 dell'Umbria, Gubbio
  - Azienda Ospedaliera di Perugia, Perugia
  - Azienda Ospedaliera di Terni, Terni

IPD SHARING:
Plan to Share IPD: Yes
IPD are available on motivated request to the principal investigator
Time Frame: 2025-2035
Access Criteria: motivated request to the principal investigator

REFERENCES:
- [Background] Bikdeli B, Caraballo C, Trujillo-Santos J, Galanaud JP, di Micco P, Rosa V, Cusido GV, Schellong S, Mellado M, Del Valle Morales M, Gavin-Sebastian O, Mazzolai L, Krumholz HM, Monreal M; RIETE Investigators. Clinical Presentation and Short- and Long-term Outcomes in Patients With Isolated Distal Deep Vein Thrombosis vs Proximal Deep Vein Thrombosis in the RIETE Registry. JAMA Cardiol. 2022 Aug 1;7(8):857-865. doi: 10.1001/jamacardio.2022.1988. PMID 35830171
- [Result] Tini G, Moriconi A, Ministrini S, Zullo V, Venanzi E, Mondovecchio G, Campanella T, Marini E, Bianchi M, Carbone F, Pirro M, De Robertis E, Pasqualini L. Ultrasound screening for asymptomatic deep vein thrombosis in critically ill patients: a pilot trial. Intern Emerg Med. 2022 Nov;17(8):2269-2277. doi: 10.1007/s11739-022-03085-8. Epub 2022 Aug 31. PMID 36044159